CLINICAL TRIAL: NCT01887795
Title: Phase Ⅲ Trial of WBRT Versus Erlotinib Concurrent Whole-brain Radiation Therapy as ﬁrst-line Treatment for Patients With Multiple Brain Metastases From Non-small-cell Lung Cancer(ENTER): a Multicentre, Open-label, Randomised Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhen-zhou Yang, Director, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yang-1970
Record Dates: First submitted 2013-06-08; First posted 2013-06-27 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Brain Metastases; Non-small-cell Lung Cancer
Keywords: Informed Consent;; Ethical Principles;; Data collection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. WBRT alone (Experimental): Selected 224 patients with multiple brain metastases from NSCLC, they will be randomized to WBRT or Erotinib concurrent WBRT. It was enough to compare the efficacy of Erotinib concurrent WBRT vs. WBRT
  Interventions: Drug: WBRT
- 2. Erlotinib concurrent WBRT (Experimental): Selected 224 patients with multiple brain metastases from NSCLC, they will be randomized to WBRT or Erotinib concurrent WBRT. It was enough to compare the efficacy of Erotinib concurrent WBRT vs. WBRT
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib
  Arms: 2. Erlotinib concurrent WBRT
Drug: WBRT
  Arms: 1. WBRT alone

SUMMARY:
1. Verify the effect of Erlotinib concurrent whole-brain radiation therapy as ﬁrst-line treatment for patients with multiple brain metastases from non-small-cell lung cancer to compare with WBRT alone.
2. Verify pre-built EGFR mutation prediction model for NSCLC brain metastases

DETAILED DESCRIPTION:
All patients will be randomized to receive WBRT or Erlotinib concurrent WBRT. Erlotinib concurrent WBRT, patients were given a loading dose of erlotinib 150mg per day for 6 days, after which all patients received erlotinib 150mg per day concurrently with WBRT. Dose reduction was allowed for intolerable adverse effects (grade ≥3) such as rash or diarrhea in 50 mg increments down from 150mg to 100 mg and then to 50 mg if needed. Radiation therapy was delivered in 2.0 Gy fractions once per day 5 days per week to a total dose of 40Gy (20 fractions). Radiation was delivered as opposed lateral 8-MV beams with a Sweden precise linear accelerator.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. the pathological diagnosis of non-small cell lung cancer and detection of pulmonary primary ARMs / sequencing EGFR mutation;
3. enhanced MRI showed brain metastases ≥ 2 or NSCLC of brain metastases after resection of residual lesions in ≥ 2 / intracranial metastases in patients with new;
4. if the previous use of EGFR-TKIs, in an WBRT synchronous Erotinib before treatment to disable EGFR-TKIs ≥ 4 weeks;
5. expected survival period over 2 months;
6. KPS score ≥ 70;
7. GPA score 0.5 - 3.5;
8. a week before randomization, bone marrow and liver and kidney function in patients with meet the following criteria:

   1. HB ≥ 100, g/L ≥ 1.5 × 109/L neutrophil and platelet ≥ 100 × 109/L;
   2. total bilirubin ≤ 1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 times the upper limit of normal;
   3. more than 1.5 times the upper limit of normal serum creatinine or creatinine clearance rate ≥ 60 ml/min, urea N ≤ 200mg/L;
   4. Urine dipstick testing the proteinuria < 1+; if the urine dipstick test value, 1+, is 24 hours total urine protein must < 500mg.
9. compliance research plan and follow-up process, and be able to carry out oral therapy;
10. in women of childbearing age, must be in before starting treatment within 7 day of urine pregnancy test and the result is negative, and not in the lactation period, and reproductive age men and women prior to entry into the study, the research process until 90 days after stopping all agree to use reliable methods of contraception;
11. can understand and consent.

Exclusion Criteria:

1. patients have been treated with radiation to the brain or to erlotinib and its ingredients allergies;
2. mixed with small cell lung cancer patients with components;
3. 5 years before other cancers except NSCLC treatment in patients with the start of the study (except for simple operation resection and there are at least 5 consecutive years disease free survival, has been cured of cervical carcinoma in situ, has cured the base cell cancer and bladder epithelial tumor);
4. before entering the group 4 weeks received any other investigational drugs;
5. judgment according to the researchers, there are serious harm to patient safety or affect the patients completed the study with the disease, and patient compliance with the difference;
6. had any clinical evidence of moderate to severe chronic obstructive pulmonary disease (COPD -COPD a history or risk factors of pulmonary function testing, FEV1/FVC<70%, FEV1<80% estimates, with or without chronic cough, sputum, difficulty breathing), activity of interstitial lung disease (-ILD pulmonary function test FEV1/FVC<70%, FEV1<80% estimates, dispersion carbon monoxide lung volume -DLCO<40%, high resolution CT showed a diffuse interstitial lung disease) disease activity and other researchers decided;
7. on gastrointestinal physiology is not perfect, or absorb the obstacle syndrome, or unable to tolerate oral medication, or active peptic ulcer;
8. any unstable system diseases: including active infection, uncontrolled hypertension, unstable angina pectoris, within the last 3 months of the onset of angina, congestive heart failure, the group in June before the myocardial infarction, need serious mental disorder drug treatment, liver, kidney or metabolic diseases; mental / spiritual diseases such as Alzheimer's disease;
9. without full control of ocular inflammation or eye infections, or any may cause the eye disease situation;
10. known human immunodeficiency virus (HIV) infection;
11. with immunodeficiency disease, or suffer from other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
12. any disease, metabolic disorders, or physical examination or laboratory suspicion or treatment of complications in patients at high risk of drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2013-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Time to neurologic progression | 13 months
  A) assess the local control of brain metastases status (including: the proportion of salvage therapy, the proportion of radiation necrosis lesions)
  B) evaluation of intracranial metastasis status (at the site of the primary tumor than the emergence of new brain metastases)

SECONDARY OUTCOMES:
Overall Survival | 3 years
Complete response, Partial response, Stable disease, Progressive disease | 19 months
Quality of Life | 3 years

OTHER OUTCOMES:
The purpose of exploring | 3 years
  1. Focal EGFR 1 certification pre built NSCLC mutation prediction model of brain metastasis.
  2. Blood sample was collected for patients with Erotinib biomarker research.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhenzhou-Yang, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Tang F, Zhang J, Xu Z, Zhang Y, Zhang X, Peng Y, Yang Z. Health-related quality of life analysis from ENTER, a randomized, controlled phase III trial of whole-brain radiotherapy with and without concurrent erlotinib in NSCLC with brain metastases. Transl Lung Cancer Res. 2024 Dec 31;13(12):3289-3302. doi: 10.21037/tlcr-24-481. Epub 2024 Dec 27. PMID 39830774
- [Derived] Yang Z, Zhang Y, Li R, Yisikandaer A, Ren B, Sun J, Li J, Chen L, Zhao R, Zhang J, Xia X, Liao Z, Carbone DP. Whole-brain radiotherapy with and without concurrent erlotinib in NSCLC with brain metastases: a multicenter, open-label, randomized, controlled phase III trial. Neuro Oncol. 2021 Jun 1;23(6):967-978. doi: 10.1093/neuonc/noaa281. PMID 33331923